CLINICAL TRIAL: NCT01885429
Title: The Effect of a Leucine 'Spike' of a Sub-optimal Protein Dose on Acute Muscle Protein Synthesis
Brief Title: Effect of Supplementing a Mixed Macronutrient Beverage With Graded Doses of Leucine on Myofibrillar Protein Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 10.32.NRC
Record Dates: First submitted 2013-04-23; First posted 2013-06-25 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Muscle Protein Synthesis
Keywords: Protein Turnover; Resistance Exercise; Whey Protein; Leucine
MeSH Terms: interventions — Diet, Protein-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Positive Control (Experimental): Group 1 (Positive(+) Control) will receive: 25g of whey protein. Positive Control
  Interventions: Dietary Supplement: Positive Control
- Negative Control (Experimental): Group 2 (Negative(-) Control) will receive: 6.25g whey. Negative Control
  Interventions: Dietary Supplement: Negative Control
- Low Protein + Low Leucine Spike (Experimental): Group 3 (Low Protein + Low Leucine Spike) will receive: 6.25g whey + low added leucine. Low Protein Low Leucine Spike
  Interventions: Dietary Supplement: Low Protein Low Leucine Spike
- Low Protein + High Leucine Spike (Experimental): Group 4 (Low Protein + High Leucine Spike) will receive: 6.25g whey + high added leucine. Low Protein High Leucine Spike
  Interventions: Dietary Supplement: Low Protein High Leucine Spike
- Low Protein + High Leucine + BCAA Spike (Experimental): Group 5 (Low Protein + High Leucine + BCAA Spike) will receive: 6.25g whey + added branched-chain amino acids. Low Protein + High Leucine + BCAA Spike
  Interventions: Dietary Supplement: Low Protein + High Leucine + BCAA Spike

INTERVENTIONS:
Dietary Supplement: Positive Control — Subject consumes 25g of whey protein following unilateral exercise
  Arms: Positive Control
Dietary Supplement: Negative Control — Subject consumes 6.25g of whey protein following unilateral exercise
  Arms: Negative Control
Dietary Supplement: Low Protein Low Leucine Spike — Subject consumes 6.25g of whey protein plus 3g of leucine following unilateral exercise
  Arms: Low Protein + Low Leucine Spike
Dietary Supplement: Low Protein High Leucine Spike — Subject consumes 6.25g of whey protein plus 5g of leucine following unilateral exercise
  Arms: Low Protein + High Leucine Spike
Dietary Supplement: Low Protein + High Leucine + BCAA Spike — Subject consumes 6.25g of whey protein plus 5g of leucine plus valine and isoleucine (BCAA) following unilateral exercise
  Arms: Low Protein + High Leucine + BCAA Spike

SUMMARY:
Muscle mass is normally maintained through the regulated balance between the processes of protein synthesis (i.e. making new muscle proteins) and protein breakdown (breaking down old muscle proteins). Proteins are composed of amino acids and we know that amino acids increase muscle protein synthesis. However, not all amino acids are the same. Essential amino acids are ones that must be consumed through food, while non-essential amino acids can be made by our body. Interestingly, the essential amino acids are all that are required to increase the rate of muscle protein synthesis. In addition, the essential amino acid leucine appears to be particularly important in regulating protein synthesis. However, how leucine is able to increase protein synthesis is not entirely understood. Previously, it has been shown that 20-25 g of high-quality protein, such as that found in milk (whey), appears to be the amount of protein that maximizes the rate of muscle protein synthesis after performing a bout of resistance exercise. Thus, we aim to measure the synthesis of new muscle proteins after ingesting different amounts of protein and amino acids. We will measure muscle protein synthesis after consumption of the beverage a participant is randomized to in a leg that has done no exercise ( ie. a rested leg) and in the other leg that has done resistance exercise. Amino acids are 'strung-together' to make protein. The 'essential' amino acids must be consumed through food because our body cannot make them, thus they are consumed when you eat protein rich foods like milk or chicken. Leucine, isoleucine, and valine are simply 3 of the 8 essential amino acids that make up dietary protein. Unlike essential amino acids, 'non-essential' amino acids may be synthesized by the body, however they are also present in protein rich foods like chicken or milk. We aim to determine if it is the leucine content found in 25 g of whey protein that is primarily responsible for maximizing muscle protein synthesis at rest and following resistance exercise. We also wish to determine how muscle genes and metabolism respond to this protocol.

DETAILED DESCRIPTION:
The processes of muscle protein synthesis (MPS) and muscle protein breakdown (MPB) occur concurrently. This constant protein turnover allows the muscle fiber to change its protein structure if loading demands or diet changes. The plasticity of skeletal muscle to respond to altered loading and contractile patterns is evidence of the capacity for remodeling that a fiber can undergo. It is quite well documented for example that mitochondrial content increases with endurance-type work. In contrast, heavier loading leads to less change in mitochondrial content but increases in myofibrillar proteins. All of the aforementioned phenotypic adaptations represent a re-patterning of the muscle's genetic expression patterns, protein translation, and processes for breakdown of existing protein structures to 'insert' the new proteins. A persistent muscle protein turnover also provides for a constant mechanism of protein 'maintenance' by removing damaged proteins and replacing them with new proteins. Damage to proteins can come about through oxidation or simply mechanical damage due to high forces during lengthening contractions. Regardless of the mechanism the balance between the processes of muscle protein synthesis (MPS) and muscle protein breakdown (MPB) will determine the net gain, loss, or no change of proteins in the myofiber.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Healthy and physically active (as determined by medical and activity questionnaire)
* 18-35 years of age
* 70-90 kg body mass
* Having given informed consent

Exclusion Criteria:

* Exhibiting health risk factors as identified on the health screening questionnaire
* Having any identified metabolic or intestinal disorders
* Tobacco use
* Aspirin use in the 4 days prior to the experimental trial
* Consumption of prescription medications or any performance enhancing agent
* Inability to endure the strenuous exercise bouts e.g. injuries
* Alcohol intake during the 48 hours prior to each of the testing days
* Currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study
* Have given blood in the last three weeks
* Verbal confirmation that they have used a substance on the WADA banned list within the last year

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in myofibrillar protein synthesis | In the first 1.5h after exercise/feeding and from 1.5-4.5h after exercise/feeding
  Myofibrillar protein synthesis will be determined by the standard precursor-product method as described previously and routinely measured and published.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada